CLINICAL TRIAL: NCT05927571
Title: An Open-Label, Multicenter, Phase Ib Trial Evaluating the Safety, Pharmacokinetics, and Activity of the Combination of Cevostamab and Elranatamab in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Activity of the Combination of Cevostamab and Elranatamab in Participants With Relapsed or Refractory Multiple Myeloma (R/R MM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43979; 2023-504657-13-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Safety Lead-In Cohort (Experimental): Participants will receive cevostamab, intravenously (IV), in combination with elranatamab, subcutaneously (SC), with step-up dosing of each drug in pre-phase following which they will receive elranatamab, at the assigned dose as a SC injection until disease progression or unacceptable toxicity. Participants will also receive cevostamab at the assigned dose as IV infusion until disease progression or unacceptable toxicity or up to 1 year on treatment, whichever occurs first.
  Interventions: Drug: Cevostamab; Drug: Elranatamab; Drug: Tocilizumab
- Dose Expansion Cohort (Combined Therapy) (Experimental): Participants will receive cevostamab, IV, in combination with elranatamab, SC, with step-up dosing in pre-phase following which they will receive elranatamab, at the assigned dose as a SC injection until disease progression or unacceptable toxicity. Participants will also receive cevostamab at the assigned dose as IV infusion until disease progression or unacceptable toxicity or up to 1 year on treatment, whichever occurs first.
  Interventions: Drug: Cevostamab; Drug: Elranatamab; Drug: Tocilizumab
- Dose Expansion Cohort (Monotherapy) (Experimental): Participants will receive elranatamab SC, with step-up dosing in pre-phase following which they will receive elranatamab, at the assigned dose as a SC injection until disease progression or unacceptable toxicity.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab solution for infusion will be administered as IV as specified in each treatment arm.
  Arms: Dose Expansion Cohort (Combined Therapy); Safety Lead-In Cohort
Drug: Elranatamab — Elranatamab solution for injection will be administered SC as specified in each treatment arm.
Drug: Tocilizumab — Tocilizumab will be used as rescue medication for participants who experience a cytokine release syndrome (CRS) event.
  Arms: Dose Expansion Cohort (Combined Therapy); Safety Lead-In Cohort

SUMMARY:
The purpose of the study is to evaluate safety and tolerability of the combination of cevostamab plus elranatamab and also determine the recommended Phase II regimen (RP2R) for the study treatment. The study consists of a safety lead-in stage, and an expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Diagnosis of R/R MM per IMWG criteria
* For female participants of childbearing potential: agreement to remain abstinent or use contraception
* For male participants: agreement to remain abstinent or use a condom

Exclusion Criteria:

* Prior treatment with cevostamab or another agent targeting fragment crystallizable receptor-like 5 (FcRH5)
* Prior treatment with elranatamab
* Prior allogeneic stem cell transplantation (SCT)
* Absolute plasma cell count exceeding 500 per milliliter (mL) or 5% of the peripheral blood white cells
* Diagnosis of Waldenström macroglobulinemia or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, skin changes (POEMS) syndrome
* Participants with known history of amyloidosis
* History of autoimmune disease
* History of confirmed progressive multifocal leukoencephalopathy
* Peripheral motor polyneuropathy of prespecified grade
* Known or suspected chronic cytomegalovirus (CMV) and/or Epstein-Barr virus (EBV) infection
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Acute or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Human immunodeficiency virus (HIV) seropositivity
* History of central nervous system (CNS) myeloma disease
* Significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From signing of informed consent up to end of study (EOS) (approximately 36 months)
  Adverse events will be reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0). The severity of CRS, immune effector cell-associated neurotoxicity syndrome (ICANS) and hemophagocytic lymphohistiocytosis (HLH) will be graded based on the American Society for Transplantation and Cellular Therapy (ASTCT) Grading Scales.
Recommended Phase II Regimen (RP2R) | Up to approximately 36 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Determined by the Investigator per International Myeloma Working Group (IMWG) Criteria | Up to approximately 36 months
Complete Response (CR)/ Stringent Complete Response (sCR) Rate as Determined by the Investigator per IMWG Criteria | Up to approximately 36 months
Rate of Very Good Partial Response (VGPR) or Better, as Determined by the Investigator per IMWG Criteria | Up to approximately 36 months
Progression-Free Survival as Determined by the Investigator per IMWG Criteria | Up to approximately 36 months
Duration of Response (DOR) as Determined by the Investigator (for Participants who Achieve a Response of Partial Response (PR) or Better) | Up to approximately 36 months
Time to First Response (for Participants who Achieve a Response of PR or Better) | Up to approximately 36 months
Time to Best Response (for Participants who Achieve a Response of PR or Better) | Up to approximately 36 months
Overall Survival (OS) | Up to approximately 36 months
Serum Concentration of Cevostamab at Specified Timepoints | Up to approximately 36 months
Serum Concentration of Elranatamab at Specified Timepoints | Up to approximately 36 months
Number of Participants with Anti-Drug Antibody (ADA) Against Cevostamab | Up to approximately 36 months
Number of Participants with ADA Against Elranatamab | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital;Haematology Clinical Trials Unit, Adelaide, South Australia
  - The Alfred Hospital, Prahan, Victoria
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- South Korea (3):
  - The Catholic University of Korea - Seoul St. Mary's Hospital (Kangnam St. Mary's Hospital), Seocho
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing